CLINICAL TRIAL: NCT06378008
Title: An 8-Week, Randomized, Controlled, Examiner-Blind, Clinical Study to Evaluate the Efficacy of a Calcium Sodium Phosphosilicate Toothpaste for the Relief of Dentin Hypersensitivity in a Population of Dentin Hypersensitivity Sufferers
Brief Title: A Clinical Study to Evaluate the Anti-Sensitivity Effect of a Calcium Sodium Phosphosilicate Toothpaste in a Population of Dentin Hypersensitivity Sufferers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300100
Record Dates: First submitted 2024-04-12; First posted 2024-04-22 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test toothpaste (Experimental): Participants will dose the toothbrush with a ribbon of toothpaste, across the full brush head and will brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening), for approximately 56 days making sure to brush the sensitive areas of the two 'test teeth' carefully first. Participants who wish to rinse after brushing will be instructed to rinse with 10 milliliter (ml) water using graduated rinsing cup provided.
  Interventions: Drug: CSPS toothpaste
- Reference toothpaste (Negative control) (Active Comparator): Participants will dose the toothbrush with a ribbon of toothpaste, across the full brush head and will brush the entire dentition thoroughly for at least 1-timed minute, twice daily (morning and evening) for approximately 56 days. Participants who wish to rinse after brushing will be instructed to rinse with 10 ml water using graduated rinsing cup provided.
  Interventions: Drug: Regular fluoride toothpaste (Crest Cavity Protection)

INTERVENTIONS:
Drug: CSPS toothpaste — Toothpaste containing 5.0% weight/weight (w/w) CSPS.
  Arms: Test toothpaste
Drug: Regular fluoride toothpaste (Crest Cavity Protection) — Regular fluoride toothpaste containing 1100 parts per million (ppm) fluoride.
  Arms: Reference toothpaste (Negative control)

SUMMARY:
The aim of this study is to confirm the clinical dentin hypersensitivity (DH) efficacy of a 5 percent (%) calcium sodium phosphosilicate (CSPS) toothpaste.

DETAILED DESCRIPTION:
This will be a single center, 8-week, randomized, controlled, examiner-blind, 2-treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected 'test teeth') clinical study to evaluate the anti-sensitivity efficacy of a 5% CSPS toothpaste in a DH population. The clinical efficacy of the 5% CSPS toothpaste (test toothpaste) will be compared with that of a reference toothpaste, a commercially available, regular fluoride toothpaste with no known anti-sensitivity properties (negative control). Sufficient participants will be screened to randomize approximately 234 participants to investigational product (approximately 117 per treatment group) and to ensure approximately 210 evaluable participants complete the entire study (approximately 105 per treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of signed and dated informed consent before any study procedures are performed.
* Participant is male or female.
* Participant is 18 to 65 years of age, inclusive, at the time of signing the informed consent.
* Participant is willing and able to comply with the study visit schedule, product usage instructions, lifestyle restrictions and other study procedures.
* Participant is in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in self-reported medical history, or upon oral examination, that would impact their safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect their ability to understand and follow study requirements.
* Screening (visit 1): Participant must have

  1. History of tooth sensitivity lasting more than six months but not more than 10 years (self-reported).
  2. Good general oral health, with a minimum of 20 natural teeth.
  3. Minimum of 2 accessible, non-adjacent teeth (incisors, canines, premolars), in different quadrants, which meet all of the following criteria:

     1. Exposed dentin due to facial/cervical erosion, abrasion or gingival recession (EAR).
     2. Modified Gingival Index (MGI) = 0 directly adjacent to the exposed dentin (that is, the test area only).
     3. Clinical mobility = 0
     4. Clinically confirmed DH to both tactile and evaporative (air) stimuli: a) Qualifying tactile threshold less than or equal to (<=) 20g. b) Qualifying Schiff sensitivity score greater than or equal to (>=) 2.
* Baseline (Visit 2, Pre-Treatment): Participant must have a minimum of two, non-adjacent accessible teeth (incisors, canines, premolars), in different quadrants, with clinically confirmed DH to both tactile and evaporative (air) stimuli at both screening (Visit 1) and baseline (Visit 2). a) Qualifying tactile threshold <= 20g at screening and baseline. b) Qualifying Schiff sensitivity score >= 2 at screening and baseline.

Exclusion Criteria:

* Participant is an employee of the investigator site directly involved in the conduct of the study, or an employee of the investigator site otherwise supervised by the investigator, or a member of their immediate family.
* Participant is an employee of the sponsor directly involved in the conduct of the study or a member of their immediate family.
* Female participant who is pregnant or intending to become pregnant during the study (self-reported).
* Female participant who is breastfeeding (self-reported).
* Participant with known or suspected intolerance or hypersensitivity to the study products, any of their stated ingredients or closely related compounds (self-reported).
* Participant with a recent history (within the last year) of alcohol or other substance abuse (self-reported).
* Participant is participating in or has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days of screening (Visit 1) or plans to participate in other studies (including non-medicinal studies) during this study.
* Participant has participated in a tooth sensitivity study within 8 weeks of screening (Visit 1).
* Participant is currently using an oral care product indicated for DH relief or care of sensitive teeth or has used an anti-sensitivity product within 8 weeks of screening (Visit 1). Participants will be required to bring their current oral care products to screening (Visit 1) for staff to verify the absence of known anti-sensitivity ingredients and sensitivity-related claims on the product packaging/label text.
* Participant takes daily doses of medications/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (for example, analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, antidepressants, mood-altering and anti-inflammatory drugs).
* Screening (Visit 1): Participant has taken antibiotics in the 2 weeks prior to screening (Visit 1).
* Baseline (Visit 2, Pre-Treatment): Participant has taken antibiotics in the 2 weeks prior to baseline (Visit 2), that is, during the acclimatization period.
* Participant takes daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* Participant requires antibiotic prophylaxis for dental procedures.
* Participant has had professional tooth de-sensitising treatment within 8 weeks of screening (Visit 1).
* Participant has had a tooth bleaching procedure within 8 weeks of screening (Visit 1).
* Participant has had dental prophylaxis within 4 weeks of screening (Visit 1).
* Participant has had treatment for periodontal disease (including surgery) within 12 months of screening (Visit 1).
* Participant has had scaling or root planning within 3 months of screening (Visit 1).
* Participant with gross periodontal disease.
* Participant with a tongue or lip piercing.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* Specific dentition exclusions for 'Test teeth':

  1. Tooth with evidence of current/recent caries.
  2. Tooth with (self-reported) treatment for decay within 12 months of screening (Visit 1).
  3. Tooth with exposed dentin and deep, defective or facial restorations.
  4. Tooth with a full crown or veneer.
  5. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or dentally qualified designee, could impact study outcomes.
  6. Sensitive tooth with contributing etiologies other than EAR to exposed dentin.
  7. Sensitive tooth not expected to benefit from use of an anti-sensitivity toothpaste, in the opinion of the investigator or dentally qualified designee.
* Participant has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Canada.
Pre-assignment Details: A total of 217 participants were screened and enrolled of which 215 participants were randomized to receive treatment in 2 groups: Test Toothpaste group (107 participants) and Reference Toothpaste group (108 participants). 2 screened participants were not randomized in the study due to other reason (scheduling issue). All randomized participants completed the study.
Groups:
- Test Toothpaste (Calcium Sodium Phosphosilicate [CSPS] Toothpaste): Participants were instructed to apply a ribbon of Test toothpaste (Toothpaste containing 5.0 percent [%] weight by weight [w/w] CSPS and 1040 parts per million [ppm] fluoride as sodium monofluorophosphate) and brush the entire dentition thoroughly for at least 1-timed minute, twice-daily (morning and evening) for approximately 56 days, making sure to brush the sensitive areas of the 2 'Test teeth' carefully first.
- Reference Toothpaste (Regular Fluoride Toothpaste): Participants were instructed to apply a ribbon of Reference toothpaste (Regular fluoride toothpaste containing 1100 ppm fluoride as sodium fluoride) and brush the entire dentition thoroughly for at least 1-timed minute, twice-daily (morning and evening) for approximately 56 days.
Period: Overall Study
Arm/Group | Test Toothpaste (Calcium Sodium Phosphosilicate [CSPS] Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Started | 107 | 108
Completed | 107 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) population included all randomized participants who received at least one dose of investigational product and completed at least one-post Baseline dentin hypersensitivity (DH) efficacy assessment.
Groups:
- Test Toothpaste (CSPS Toothpaste): Participants were instructed to apply a ribbon of Test toothpaste (Toothpaste containing 5% w/w CSPS and 1040 ppm fluoride as sodium monofluorophosphate) and brush the entire dentition thoroughly for at least 1-timed minute, twice-daily (morning and evening) for approximately 56 days, making sure to brush the sensitive areas of the 2 'Test teeth' carefully first.
- Total: Total of all reporting groups
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste) | Total
Number analyzed (Participants) | 107 | 108 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (13.53) | 50.4 (12.76) | 48.4 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 75 | 147
  Male | 35 | 33 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 104 | 103 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 48 | 29 | 77
  Asian - Central/South Asian Heritage | 4 | 4 | 8
  Asian - East Asian Heritage | 4 | 3 | 7
  Asian - South East Asian Heritage | 8 | 7 | 15
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 41 | 64 | 105
  Multiple | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score at Day 56
Description: Evaporative (air) sensitivity was assessed on facial surfaces of teeth by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface. Participant's response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative (air) stimulus. Score ranged from 0-3, where 0=Did not respond to air stimulation; 1=Responded to air stimulus but did not request discontinuation of stimulus; 2=Responded to air stimulus and requested discontinuation or moved from stimulus; 3=Responded to stimulus, considered stimulus to be painful, requested discontinuation of the stimulus. Schiff sensitivity score = Mean score for the two 'Test Teeth' selected at Baseline by the examiner. Lower score=low degree of sensitivity. Change from Baseline (Day 0) was calculated by subtracting Baseline score from Day 56 score. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) and Day 56
Population: mITT population included all randomized participants who received at least one dose of investigational product and completed at least one-post Baseline DH efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale | -2.00 (0.065) | -0.20 (0.065)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.80, 95% CI 2-sided [-1.98 to -1.62], Standard Error of Mean 0.092 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste

2. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold (Gram [g]) at Day 56
Description: Tactile sensitivity was assessed for the 2 test teeth selected at Baseline by the examiner using a constant pressure probe (Yeaple probe). The probe tip was placed perpendicular to the facial surface of tooth and drawn slowly across the exposed dentine. After each application, the participants were asked to indicate whether they experienced any pain or discomfort (yes/no response). The gram setting with two consecutive 'yes' responses was recorded as the tactile threshold in gram for that tooth. At Baseline, the upper force setting was 20 g. Tactile threshold (g) was derived as the mean value for the 2 'Test Teeth' selected at Baseline by the examiner. Higher tactile threshold indicated less sensitivity. Change from Baseline was calculated by subtracting Baseline (Day 0) value from Day 56 value. A positive change from Baseline indicated improvement.
Time Frame: Baseline (Day 0) and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
grams | 56.79 (1.721) | 3.92 (1.713)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 52.87, 95% CI 2-sided [48.08 to 57.65], Standard Error of Mean 2.428 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste

3. Secondary Outcome: Adjusted Mean Change From Baseline in Schiff Sensitivity Score at Days 3, 7, 14 and 28
Description: Evaporative(air) sensitivity was assessed on facial surfaces of teeth by directing a 1 second application of air from standard dental syringe held perpendicular to tooth surface. Participant's response to the stimulus was evaluated using the Schiff sensitivity scale, an examiner-based index scored immediately following administration of the evaporative(air) stimulus. Score ranged from 0-3, where 0=Did not respond to air stimulation;1=Responded to air stimulus but did not request discontinuation of stimulus;2=Responded to air stimulus and requested discontinuation or moved from stimulus;3=Responded to stimulus, considered stimulus to be painful, requested discontinuation of the stimulus. Schiff sensitivity score=Mean score for the 2 'Test Teeth' selected at Baseline by examiner. Lower score=low degree of sensitivity. Change from Baseline was calculated by subtracting the Baseline(Day 0) score from score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Days 3, 7, 14 and 28
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 3 | -0.31 (0.038) | -0.12 (0.038)
  Change from Baseline at Day 7 | -0.73 (0.045) | -0.12 (0.045)
  Change from Baseline at Day 14 | -1.37 (0.065) | -0.14 (0.065)
  Change from Baseline at Day 28 | -1.76 (0.066) | -0.20 (0.066)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 3; Test type: Superiority; p = 0.0005, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.19, 95% CI 2-sided [-0.29 to -0.08], Standard Error of Mean 0.053 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 7; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.61, 95% CI 2-sided [-0.73 to -0.49], Standard Error of Mean 0.063 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 3: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.23, 95% CI 2-sided [-1.41 to -1.04], Standard Error of Mean 0.092 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 4: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.56, 95% CI 2-sided [-1.74 to -1.38], Standard Error of Mean 0.093 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste

4. Secondary Outcome: Adjusted Mean Change From Baseline in Tactile Threshold (g) at Days 3, 7, 14 and 28
Description: as for outcome 2
Time Frame: Baseline (Day 0), Days 3, 7, 14 and 28
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
grams
  Change from Baseline at Day 3 | 8.05 (0.500) | 0.91 (0.497)
  Change from Baseline at Day 7 | 16.79 (0.788) | 2.39 (0.784)
  Change from Baseline at Day 14 | 28.56 (1.127) | 2.76 (1.121)
  Change from Baseline at Day 28 | 44.08 (1.597) | 3.09 (1.590)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 7.14, 95% CI 2-sided [5.75 to 8.53], Standard Error of Mean 0.706 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 7; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 14.40, 95% CI 2-sided [12.20 to 16.59], Standard Error of Mean 1.112 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 3: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 14; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 25.80, 95% CI 2-sided [22.67 to 28.93], Standard Error of Mean 1.590 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste
Statistical Analysis 4: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = 40.99, 95% CI 2-sided [36.55 to 45.43], Standard Error of Mean 2.254 — Adjusted mean difference was calculated as test toothpaste minus reference toothpaste

5. Secondary Outcome: Adjusted Mean Change From Baseline in Impact on Everyday Life (Section 1 of Dentin Hypersensitivity Experience Questionnaire [DHEQ-48], Question [Q]7-9) at Days 28 and 56
Description: The DHEQ is a validated, condition-specific measure of Oral Health-Related Quality of Life (OHRQoL) in relation to DH. DHEQ Section 1, questions 7-9 were about participant's sensitive teeth and its impact on their everyday life. Participants scored Q7 (how intense are the sensations?) on a scale of 1 (not at all intense) to 10 (worst imaginable); Q8 (how bothered are you by any sensations?) on a scale of 1 (not at all bothered) to 10 (extremely bothered); Q9 (how well can you tolerate sensations?) on a scale of 1 (can easily tolerate) to 10 (can't tolerate at all). The total score for each question ranged from 1 to 10; where lower score indicated less intense, less bothersome and tolerable sensations. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Q7 (How intense are the sensations?): Change from Baseline at Day 28 | -0.60 (0.167) | -0.26 (0.143)
  Q7 (How intense are the sensations?): Change from Baseline at Day 56 | -0.77 (0.213) | -0.18 (0.161)
  Q8 (How bothered are you by any sensations?): Change from Baseline at Day 28 | -0.63 (0.196) | -0.53 (0.159)
  Q8 (How bothered are you by any sensations?): Change from Baseline at Day 56 | -0.86 (0.222) | -0.54 (0.173)
  Q9 (How well can you tolerate sensations?): Change from Baseline at Day 28 | -0.45 (0.202) | -0.29 (0.166)
  Q9 (How well can you tolerate sensations?): Change from Baseline at Day 56 | -0.63 (0.206) | 0.18 (0.211)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q7 (How intense are the sensations?): Change from Baseline at Day 28; Test type: Superiority; p = 0.3489, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.21, 95% CI 2-sided [-0.64 to 0.23], Standard Error of Mean 0.219 — Adjusted Mean Difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q7 (How intense are the sensations?): Change from Baseline at Day 56; Test type: Superiority; p = 0.0876, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.46, 95% CI 2-sided [-0.98 to 0.07], Standard Error of Mean 0.267 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 3: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q8 (How bothered are you by any sensations?): Change from Baseline at Day 28; Test type: Superiority; p = 0.9108, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.03, 95% CI 2-sided [-0.47 to 0.52], Standard Error of Mean 0.252 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 4: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q8 (How bothered are you by any sensations?): Change from Baseline at Day 56; Test type: Superiority; p = 0.4854, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.20, 95% CI 2-sided [-0.75 to 0.36], Standard Error of Mean 0.281 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 5: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q9 (How well can you tolerate sensations?): Change from Baseline at Day 28; Test type: Superiority; p = 0.8309, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.06, 95% CI 2-sided [-0.46 to 0.57], Standard Error of Mean 0.261 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 6: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Q9 (How well can you tolerate sensations?): Change from Baseline at Day 56; Test type: Superiority; p = 0.0500, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.58, 95% CI 2-sided [-1.17 to -0.00], Standard Error of Mean 0.297 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

6. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Total Score (Section 2, Question Q1-34) at Days 28 and 56
Description: DHEQ is a validated, condition-specific measure of OHRQoL in relation to DH. Section 2 of DHEQ included 34 questions grouped into 5 domains: Restrictions(Q1-4), Adaptation(Q5-16), Social Impact(Q17-21), Emotional Impact(Q22-29), and Identity(Q30-34). Participants scored each question using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score was derived as sum of all questions (Q1 to Q34) score and ranged from 34 to 238, where lower score indicated better OHrQoL. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from the score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -5.77 (2.756) | -3.22 (2.689)
  Change from Baseline at Day 56 | -18.71 (3.465) | -12.48 (3.205)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.5565, Mixed Model with Repeated Measures; Adjusted Mean Difference = -2.27, 95% CI 2-sided [-9.88 to 5.33], Standard Error of Mean 3.859 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.2078, Mixed Model with Repeated Measures; Adjusted Mean Difference = -5.96, 95% CI 2-sided [-15.25 to 3.34], Standard Error of Mean 4.715 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

7. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Restrictions Domain (Section 2, Q1-4) Score at Days 28 and 56
Description: Restrictions domain of DHEQ evaluated the ways in which any sensations in participant's teeth affected them in their daily life. It included 4 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 4 to 28. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from the score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -0.87 (0.367) | 0.05 (0.452)
  Change from Baseline at Day 56 | -2.82 (0.503) | -1.73 (0.491)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.5597, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.34, 95% CI 2-sided [-1.50 to 0.82], Standard Error of Mean 0.588 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.4627, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.52, 95% CI 2-sided [-1.91 to 0.87], Standard Error of Mean 0.705 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

8. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Adaptation Domain Score (Section 2, Q5-16) at Days 28 and 56
Description: Adaptation domain of DHEQ evaluated 'the ways in which the sensations in participant's teeth had forced them to change things in their daily life', 'things they did in their daily life to avoid experiencing the sensations in their teeth'. It included 12 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 12 to 84. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from the score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -2.71 (1.176) | -0.57 (1.059)
  Change from Baseline at Day 56 | -7.49 (1.473) | -4.46 (1.294)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.3000, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.64, 95% CI 2-sided [-4.77 to 1.48], Standard Error of Mean 1.583 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.1974, Mixed Model with Repeated Measures; Adjusted Mean Difference = -2.53, 95% CI 2-sided [-6.39 to 1.33], Standard Error of Mean 1.958 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

9. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Social Impact Domain (Section 2, Q17-21) Score at Days 28 and 56
Description: Social Impact domain of DHEQ evaluated the way the sensations affected participants when they were with other people or in certain situations. It included 5 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 5 to 35. Lower score indicated less effect of sensations on participant's social life. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from the score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -0.23 (0.454) | -0.36 (0.503)
  Change from Baseline at Day 56 | -2.18 (0.533) | -1.41 (0.480)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.9203, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.07, 95% CI 2-sided [-1.27 to 1.41], Standard Error of Mean 0.679 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.2489, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.83, 95% CI 2-sided [-2.24 to 0.58], Standard Error of Mean 0.717 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

10. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Emotional Impact Domain (Section 2, Q22-29) Score at Days 28 and 56
Description: Emotional Impact domain of DHEQ evaluated the way the sensations in participant's teeth made them feel. It included 8 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 8 to 56. Lower score indicated less effect of sensations on participant's emotions. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from the score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -1.52 (0.794) | -1.54 (0.743)
  Change from Baseline at Day 56 | -5.02 (0.918) | -3.51 (0.820)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.8496, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.21, 95% CI 2-sided [-2.36 to 1.94], Standard Error of Mean 1.090 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.1596, Mixed Model with Repeated Measures; Adjusted Mean Difference = -1.73, 95% CI 2-sided [-4.15 to 0.69], Standard Error of Mean 1.226 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

11. Secondary Outcome: Adjusted Mean Change From Baseline in DHEQ Identity Domain (Section 2, Q30-34) Score at Days 28 and 56
Description: Identity domain of DHEQ evaluated what the sensations in participant's teeth meant for them. It included 5 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 5 to 35, where lower score indicated less impact of sensations on participant's identity. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -0.43 (0.509) | -0.80 (0.475)
  Change from Baseline at Day 56 | -1.21 (0.568) | -1.37 (0.489)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.9577, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.04, 95% CI 2-sided [-1.34 to 1.41], Standard Error of Mean 0.697 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.8261, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.16, 95% CI 2-sided [-1.64 to 1.31], Standard Error of Mean 0.748 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

12. Secondary Outcome: Adjusted Mean Change From Baseline in Global Oral Health (DHEQ Section 2, Q35) Score at Days 28 and 56
Description: Global Oral Health was evaluated using a single question of DHEQ about overall health of participant's mouth, teeth, and gums. Participants rated the overall health of their mouth, teeth, and gums using a 6-point scale ranging from 1 to 6 where 1=excellent, 2=very good, 3=good, 4=fair, 5=poor, and 6=very poor. Lower score indicated better oral health. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from score at each indicated timepoint. A negative change from Baseline indicated improvement.
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -0.06 (0.070) | -0.06 (0.055)
  Change from Baseline at Day 56 | -0.07 (0.070) | -0.10 (0.072)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.8895, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.01, 95% CI 2-sided [-0.19 to 0.16], Standard Error of Mean 0.089 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.8083, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.02, 95% CI 2-sided [-0.17 to 0.22], Standard Error of Mean 0.101 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

13. Secondary Outcome: Adjusted Mean Change From Baseline in Effect on Life Overall (DHEQ Section 2, Q36-39) Score at Days 28 and 56
Description: Effect on Life was evaluated using 4 questions about how much the sensations in teeth affected participant's life overall. Participants scored each question on a 5-point scale ranging from 0 to 4 where 0=not at all, 1=a little, 2=somewhat; 3=quite a bit, and 4=very much. Thus, the total score ranged from 0 to 16, where lower score indicated less impact of sensations on participant's life overall. Change from Baseline was calculated by subtracting the Baseline (Day 0) score from score at each indicated timepoint. A negative change from Baseline indicated improvement
Time Frame: Baseline (Day 0), Day 28 and Day 56
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
Number analyzed (Participants) | 107 | 108
score on a scale
  Change from Baseline at Day 28 | -0.45 (0.272) | -0.63 (0.225)
  Change from Baseline at Day 56 | -1.04 (0.303) | -0.87 (0.247)
Statistical Analysis 1: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 28; Test type: Superiority; p = 0.7362, Mixed Model with Repeated Measures; Adjusted Mean Difference = 0.12, 95% CI 2-sided [-0.57 to 0.81], Standard Error of Mean 0.351 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste
Statistical Analysis 2: Comparison: Test Toothpaste (CSPS Toothpaste) vs Reference Toothpaste (Regular Fluoride Toothpaste); Change from Baseline at Day 56; Test type: Superiority; p = 0.5568, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.23, 95% CI 2-sided [-1.00 to 0.54], Standard Error of Mean 0.390 — Adjusted mean difference was calculated as Test Toothpaste minus Reference Toothpaste

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product (or the last study procedure) (up to approximately 90 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including an acclimatization product (or medical device), whether or not considered related to the study product, including an acclimatization product (or medical device). A serious adverse event (SAE) was a particular category of AE where the adverse outcome was serious.
Arm/Group | Test Toothpaste (CSPS Toothpaste) | Reference Toothpaste (Regular Fluoride Toothpaste)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/108
Other Adverse Events (participants affected / at risk) | 0/107 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT06378008/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06378008/SAP_001.pdf